CLINICAL TRIAL: NCT01292174
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Sequential Dose-Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered Ibalizumab in HIV-Negative, At-Risk Volunteers
Brief Title: Safety Study of Ibalizumab Subcutaneous Injection in Healthy Volunteers
Acronym: TMB-108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Collaborators: Aaron Diamond AIDS Research Center (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TMB-108
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Prevention of Infection With HIV-1
Keywords: HIV prevention
MeSH Terms: interventions — ibalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 - lowest dosage (Experimental): 120 mg ibalizumab administered by subcutaneous injection weekly for 4 weeks, randomized 6:2 with placebo
  Interventions: Biological: ibalizumab (biologic/MAb) for SC Injection or placebo
- Group 2 - middle dosage level (Experimental): 240 mg ibalizumab administered by subcutaneous injection weekly for 4 weeks, randomized 6:2 with placebo
  Interventions: Biological: ibalizumab (biologic/MAb) for SC Injection or placebo
- Group 3 - highest dosage level (Experimental): 480 mg ibalizumab administered by subcutaneous injection weekly for 4 weeks, randomized 6:2 with placebo
  Interventions: Biological: ibalizumab (biologic/MAb) for SC Injection or placebo

INTERVENTIONS:
Biological: ibalizumab (biologic/MAb) for SC Injection or placebo — ibalizumab or matching placebo administered by subcutaneous injection weekly at 120 mg
  Other Names: formerly TNX-355
  Arms: Group 1 - lowest dosage
Biological: ibalizumab (biologic/MAb) for SC Injection or placebo — ibalizumab or matching placebo administered by subcutaneous injection weekly at 240 mg
  Other Names: formerly TNX-355
  Arms: Group 2 - middle dosage level
Biological: ibalizumab (biologic/MAb) for SC Injection or placebo — ibalizumab or matching placebo administered by subcutaneous injection weekly at 480 mg
  Other Names: formerly TNX-355
  Arms: Group 3 - highest dosage level

SUMMARY:
The is a blinded safety study of ibalizumab given by subcutaneous injection in sequentially increasing dose-groups of at-risk, HIV-negative, healthy volunteers. The study involves the administration of four total injections of ibalizumab or matching placebo in each volunteer, given once every week, at one of three dose levels. Drug administration begins at the lowest dose. After 4 of 8 volunteers in the first group have received all study drug injections and have completed 6 additional weeks of follow-up, an independent safety monitoring group will review available data before approving initiation of the next higher dose-group. This process will be repeated prior to initiation of the 3rd and highest dose-group.

All volunteers will participate in 2 separate intensive blood sampling periods of 7 days each to test drug levels.

DETAILED DESCRIPTION:
The study is a phase 1, randomized, double-blinded, placebo-controlled, sequential dose-escalation and safety study of ibalizumab in at-risk HIV-negative volunteers. The study involves the administration of four total injections of ibalizumab or matching placebo in each volunteer, given once every week, in one of three groups as defined below:

Group 1: 120 mg sc weekly x 4 weeks, randomized 6:2 with placebo Group 2: 240 mg sc weekly x 4 weeks, randomized 6:2 with placebo Group 3: 480 mg sc weekly x 4 weeks, randomized 6:2 with placebo

Volunteers will be screened up to 42 days prior to enrollment and first drug administration, and will be followed for 26 weeks after the final injection.

All subjects will be expected to participate in two (2) intense PK sampling periods with a duration of 7 days for the first period and 14 days for the second period. During these periods (following Day 0 and following Week 3) subjects will have daily serum concentration and other investigational pharmacokinetic assessments.

All volunteers will be encouraged to participate in an optional collection of genital secretions (semen or vaginal wash) at Week 4.

An independent data safety monitoring board (DSMB) will review study data after four out of eight at-risk HIV-negative volunteers in Group 1 (120 mg dose) have received all study drug injections and completed 6 weeks of follow-up before approving escalation to Group 2 (240 mg dose). The DSMB will also review all available study data from Groups 1, and 2 after four out of eight volunteers in Group 2 have received all study drug injections and completed 6 weeks of follow-up before approving escalation to Group 3 (480 mg dose).

ELIGIBILITY:
Inclusion Criteria:

1. At-risk adult males and females, as assessed by a medical history, physical exam, and laboratory tests
2. At least 18 years of age and no greater than 40 years on the day of screening
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study
4. In the opinion of the principal investigator or designee, has understood the information provided; written informed consent needs to be given before any study-related procedures are performed
5. Willing to undergo HIV Testing and counseling, and receive HIV test results
6. Agrees to use a barrier form of contraception if engaging in sexual activity at any time throughout the study and the follow-up period (males and females) - two reliable forms of contraception, one barrier and one hormonal (e.g., oral contraceptive pill, injectable or implantable contraceptive combined with diaphragm, Intra Uterine Device (IUD), or condoms), must be used if volunteers engage in sexual activity that could result in pregnancy; is anatomically sterile in self or partner; all female volunteers must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Events and Procedures

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the trial physician within the last 6 months
3. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
4. Any laboratory value of Grade 1 or higher according to the NCI Common Toxicity Criteria
5. Confirmed diagnosis of hepatitis B (surface antigen, HbsAg) or hepatitis C (HCV antibodies)
6. Current confirmed STD infection
7. Prior receipt of Hepatitis A vaccine by history, or anti-hepatitis A antibodies at screening
8. Pregnant, planning a pregnancy during the trial period, or lactating
9. Receipt of a live attenuated vaccine (other than influenza) within 30 days or other vaccine within 14 days of study enrollment
10. Receipt of blood transfusion or blood products 6 months prior to study drug administration
11. Participation in another clinical study of an investigational product currently or within 30 days prior to Screening, or expected participation during this study
12. History of severe allergic reactions or known allergy to any component of the study drug
13. Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, suicide attempt in the previous 3 years
14. In the opinion of the investigator, unlikely to comply with protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of subcutaneous administration of ibalizumab in at-risk HIV-negative volunteers | 30 weeks
  Safety and Tolerability Measures Include:
  * Physical examinations
  * Vital sign measurements
  * Anti-ibalizumab antibody levels (immunogenicity of ibalizumab)
  * Clinical laboratory parameters (hematology, serum chemistry and urinalysis)
  * Urine or serum pregnancy tests
  * Adverse events
  * Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Stanley T Lewis, MD, MPH, Study Director — TaiMed Biologics, USA
Locations (6):
- United States (6):
  - Alabama Vaccine Research Center, Birmingham, Alabama
  - Living Hope Clinical Foundation, Long Beach, California
  - Quest Clinical Research, San Francisco, California
  - ACRIA - AIDS Community Research Initiative of America, New York, New York
  - University of Rochester, Rochester, New York
  - Research Access Network / The Schrader Clinic, Houston, Texas